CLINICAL TRIAL: NCT00131430
Title: An 18-Month Study to Assess the Safety, Tolerability, and Efficacy of MK0364 in Obese Patients
Brief Title: An Eighteen Month Efficacy and Safety Study in Obese Patients (0364-020)(COMPLETED)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0364-020; 2005_044; MK-0364-020
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-03

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: taranabant
  Other Names: MK0364

SUMMARY:
A study to determine the safety and efficacy of an investigational drug in patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with a body mass index between 30kg/m2 and 43 kg/m2, inclusive (BMI between 27 kg/m2 and 43kg/m2, inclusive for those with obesity-related comorbidities including hypertension, dyslipidemia and sleep apnea).

Exclusion Criteria:

* Patients with serious or unstable current or past medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
After 24 weeks, body weight, safety, and tolerability | After 24 weeks

SECONDARY OUTCOMES:
After 80 weeks, body weight | After 80 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC